CLINICAL TRIAL: NCT05877846
Title: A Precision Nutrition Approach to Enhancing Physical Function in Older Adults: A Pilot, Feasibility Study
Brief Title: Precision Medicine and Physical Function
Acronym: HMB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-0141
Record Dates: First submitted 2023-05-10; First posted 2023-05-26 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Frailty; Weakness, Muscle; Multiple Chronic Conditions
MeSH Terms: conditions — Frailty; Muscle Weakness; Multiple Chronic Conditions | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: This pilot study is a 12-week, single arm, pre/post intervention of β-hydroxymethyl butyrate (HMB) in n=18 older adults at risk for sarcopenia. There will be no randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Weakness (Experimental): Participants will take beta-hydroxymethyl butyrate (HMB) with vitamin D3 for 12 weeks. Those participants with vitamin D3 levels > 80 ng/dL will be provided intervention capsules without vitamin D3.
  Interventions: Dietary Supplement: Beta-hydroxymethyl butyrate supplement; Dietary Supplement: Vitamin D supplement; Dietary Supplement: Matching Beta-hydroxymethyl butyrate supplement without Vitamin D

INTERVENTIONS:
Dietary Supplement: Beta-hydroxymethyl butyrate supplement — Beta-hydroxymethyl butyrate (750 mg) - Vitamin D3 (200 IU) capsules. The formulation is 750 mg of Beta-hydroxymethyl butyrate with 200 IU of vitamin D3 per capsule. Frequency is 2 capsules twice daily (morning, evening)
Dietary Supplement: Vitamin D supplement — Beta-hydroxymethyl butyrate (750 mg) - Vitamin D3 (200 IU) capsules. The formulation is 750 mg of Beta-hydroxymethyl butyrate with 200 IU of vitamin D3 per capsule. Frequency is 2 capsules twice daily (morning, evening)
Dietary Supplement: Matching Beta-hydroxymethyl butyrate supplement without Vitamin D — Beta-hydroxymethyl butyrate (750 mg) capsules. The formulation is 750 mg of Beta-hydroxymethyl butyrate per capsule. Frequency is 2 capsules twice daily (morning, evening)

SUMMARY:
The investigators aim to conduct a 12-week, single-arm, pre/post-intervention of b-hydroxy-methylbutyrate in persons aged 65 to 85 years to assess feasibility and acceptability of the intervention and study procedures, secondary outcomes of physical function and changes in multi-omics patterns, and exploratory outcomes that will allow the team to describe physical function phenotype. The investigators' primary outcomes are the: feasibility of the study procedures (including safety), feasibility of the intervention delivery, and acceptability of study procedures and measures. Secondary outcomes include: Objective and subjective physical function measures that predict disability including the 30-second sit-to-stand, knee strength, isokinetic strength, grip strength, gait speed, 400-m walk test, Pittsburgh Fatiguability, PROMIS global health-10, social support, anthropometry, National Institutes of Health (NIH) Cognitive toolbox, Automated Self-Administered 24-hour Dietary Assessment (ASA-24), Community Healthy Activities Model Programs (CHAMPS), Ultrasound Imaging, Magnetic Resonance Imaging (MRI), Changes in untargeted metabolomic profile data based on qualitative or semiquantitative analysis of the most probable detectable metabolites in laboratory samples , Discover potential metabolites that explain changes in physical function using a discovery science, precision medicine approach (discovery science approach that is exploratory)

ELIGIBILITY:
Inclusion Criteria:

* English-speaking older adults aged 65 to 85 years (of all genders and sexes, race or ethnicity)
* A University of North Carolina at Chapel Hill (UNC) Geriatrics Medicine clinic patient;
* Chronic medical conditions -these are based on the 21 Medicare multiple chronic conditions (e.g., alcohol abuse, arthritis (osteoarthritis, rheumatoid), asthma, atrial fibrillation, autism spectrum disorders, cancer (breast, colorectal, lung, prostate), chronic kidney disease, chronic obstructive pulmonary disease, depression, diabetes, drug/substance abuse, heart failure, hepatitis, HIV/AIDS, hyperlipidemia, hypertension, ischemic heart disease, osteoporosis, schizophrenia/other psychotic disorders, stroke);

Exclusion Criteria:

* Age <65 years and >85 years old
* A medical diagnosis of dementia
* Those without a negative subjective weakness screener (<1)
* Individuals with life-threatening or untreated psychiatric diagnosis that would interfere with study participation and require significant modification to meet their needs such as untreated major depressive disorder, substance abuse, suicidal ideation or untreated severe mental illness (schizophrenia, bipolar disorder)
* Life-threatening illness including those receiving palliative care or hospice services
* Individuals unwilling/unable to provide consent
* Inability to complete the protocol procedures
* Elective surgery in the next four months
* Medications - antiobesity (weight loss agents) medications that lead to weight loss
* Hospitalization for heart failure in past 6 months, advanced non-skin cancer (Stage III or IV) on treatment; Advanced liver failure; Chronic renal insufficiency on hemodialysis; advanced Chronic obstructive pulmonary disease (COPD) that would prevent engagement

  ***Vitamin D >80 ng/dL:
* At baseline, the investigators will check Vit D levels - recognize that processing is highly dependent on the McLendon lab and may take up to 7+ days to come back.
* Concurrently, the investigators will consider continuing consent, enrollment, study procedures.
* Provide at Visit 2 the beta-hydroxymethyl butyrate/Vitamin D supplement
* Once the results have been received and reviewed - if the levels exceed 80 ng/dL, then the participant will be informed.
* At that point, the investigators will either exclude the participant or, if available, see whether the company is willing to provide formulations of just beta-hydroxymethyl butyrate (HMB)and provide this to the participant
* These guidelines account for the fact that Vit D is not recommended by American Geriatrics Society to check routinely, and that levels <80 (or even 120 ng/mL) rarely lead to toxicity.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Enrolled | at 12-weeks
  Feasibility of study procedures is measured by the percentage of enrolled participants that were screened (percent participants enrolled = number of participants enrolled/number of participants screened x 100). There are no cut-off scores for interpretation but, higher scores indicate greater feasibility of the study.
Number of Participants Screened | Through the end of the study period (~1 year) based on data collected on each participant at the conclusion of the study intervention (12-weeks).
  Feasibility of study procedures as measured by the number of participants that were screened.
Percentage of participants consented | Through the end of the study period (~1 year) based on data collected on each participant at the conclusion of the study intervention (12-weeks).
  The percent of participants that consented in the study is defined as the number of participants that were consented divided by the # of participants screened multiplied by 100. There are no cut-off scores for interpretation but, higher scores indicate greater feasibility of the study.
Percent attendance | Through the end of the study period (~1 year) based on data collected on each participant at the conclusion of the study intervention (12-weeks).
  Feasibility of study procedures measured as the mean attendance rate of all participants. Participant attendance rate = (total # of visits attended / total # of visits scheduled) x 100. There are no cut-off scores for interpretation. Higher scores indicate higher feasibility
Percent of Interviews completed | Through the end of the study period (~1 year) based on data collected on each participant at the conclusion of the study intervention (12-weeks).
  Feasibility of study procedures measures as interview completion rate. Percent of completed interviews = (# of completed interviews / # of participants completing the intervention) x 100. There are no cut-off scores for interpretation. Higher rates are indicative of higher feasibility.
Percentage of study measures collected | 12 weeks after baseline visit
  Rate of the percent of study measures collected, defined as the # of study procedures collected divided by the total # of proposed study procedures x 100. A higher number is characteristic of increased feasibility of collecting study measures.
Percent of participants conducted MRI measure | 12 weeks after baseline visit
  Rate of participants who conducted two MRI measures, defined as the total number of MRI measures collected divided by the total expected number of MRI measures. A higher number indicates feasibility of obtaining MRI measures.
Percent of participants conducted ultrasound measure | 12 weeks after baseline visit
  Rate of participants who conducted three ultrasound measures, defined as the total number of MRI measures collected divided by the total expected number of ultrasound measures. A higher number indicates feasibility of obtaining ultrasound measures.
Acceptability of study intervention | 12 weeks after baseline visit
  Measured through an end of study satisfaction survey, acceptability is measured on a 10 point Likert scale conducted on all participants at 12-weeks. This is rated on a 1 (strongly disagree) to 10 (strongly agree) survey.
Percent of Participants Rating the Intervention as Acceptable | 12 weeks after baseline visit
  Conducted on all participants using a 1-5 Likert scale to assess appropriateness of the study intervention measures using the following: completely disagree, disagree, neither agree or disagree, agree, completely agree. Acceptability is reported as Agree or Completely Agree responses. Rate is calculated as total number of participants rating as agree or complete agree divided by the number of total participants.
Percent of participants rating the intervention as appropriate | 12 weeks after baseline visit
  Conducted on all participants using a 1-5 Likert scale to assess appropriateness of the study intervention measures using the following: completely disagree, disagree, neither agree or disagree, agree, completely agree. Intervention appropriateness is reported as Agree or Completely Agree responses. Rate is calculated as total number of participants rating as agree or complete agree divided by the number of total participants.
Percent of participants rating the intervention as feasible | 12 weeks after baseline visit
  Conducted on all participants using a 1-5 Likert scale to assess feasibility of the study intervention measures using the following: completely disagree, disagree, neither agree or disagree, agree, completely agree. Intervention feasibility is reported as Agree or Completely Agree responses. Rate is calculated as total number of participants rating as agree or complete agree divided by the number of total participants.

SECONDARY OUTCOMES:
Change in weight from baseline | At baseline, 6 weeks, and 12 weeks
  Absolute change in weight in kilograms (kg) over time from baseline to 12-weeks. Weight will be objectively measured on a digital scale. A negative number will indicate weight loss.
Change in waist circumference from baseline | At baseline, 6 weeks, and 12 weeks
  Absolute change in waist circumference in centimeters (cm) over time from baseline to 12-weeks. Waist circumference will be measured objectively using a tape measure. A negative number will indicate a loss in waist circumference
Change in hip circumference from baseline | At baseline, 6 weeks, and 12 weeks
  Absolute change in hip circumference in centimeters (cm) over time from baseline to 12-weeks. Hip circumference will be measured objectively using a tape measure. A negative number will indicate a loss of hip circumference
Change in arm circumference from baseline | At baseline, 6 weeks, and 12 weeks
  Change in arm circumference in centimeters (cm) over time from baseline to 12-weeks. Arm circumference will be measured objectively using a tape measure. A negative number will indicate a loss in arm circumference.
Change in calf circumference from baseline | At baseline, 6 weeks, and 12 weeks
  Change in calf circumference in centimeters (cm) over time from baseline to 12-weeks. Calf circumference will be measured objectively using a tape measure. A negative number will indicate a loss in calf circumference
Change in Language using the Picture Vocabulary Test | At baseline, 6 weeks, and 12 weeks
  Part of the NIH Cognitive Toolbox, Language will be measured with respondents selecting the picture that closely matches the meaning of the word. A set of mental processes that translate thought into symbols (words, gestures) that can be shared among individuals for purposes of communication. A change will be measured. This takes 4 minutes to administer. The number of items presented depends on age and performance; for most, it will contain ~25 items. The computer will administer each item one by one, in an untimed fashion, until the test is completed. The test uses age (for participants younger than 18) and education (for participants 18 and older) to determine which items it initially presents. Item Response Theory (IRT) is used to score the Picture Vocabulary Test (TPVT) which is then converted to a standardized score. Fully Corrected Score for which the normative mean is 50 and the standard deviation (SD) is 10.
Change in Executive function using the Dimensional Change Card Sort Test | At baseline, 6 weeks, and 12 weeks
  Executive Function measures the capacity to plan, organize, and monitor the execution of behaviors that are strategically directed in a goal-oriented manner. Set shifting, or the capacity for switching among multiple aspects of a strategy or task. A change will be measured. This takes 4 minutes. Two target pictures are presented that vary along two dimensions (e.g., shape and color). Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape). There are a maximum of 8 items. Unadjusted score ranges 0-40. Fully Corrected Score for which the normative mean is 50 and the standard deviation (SD) is 10. Higher scores are better cognition. A positive change is improvement in function
Change in Episodic memory using the Picture sequence memory test | At baseline, 6 weeks, and 12 weeks
  Episodic memory are cognitive processes involved in acquiring, storing, and retrieving new information. A change will be measured. This takes 7 minutes. In this measure , sequences of pictured objects and activities are presented in a particular order. The participants are asked to reproduce the sequence of pictures that is shown on the screen. Participants are given credit for each adjacent pair of pictures they correctly place (i.e., if pictures in locations 7 and 8 are placed in that order and adjacent to each other anywhere, such as slots 1 and 2, one point is awarded), up to the maximum value for the sequence, which is one less than the sequence length. (That is, if 18 pictures are in the sequence, the maximum score on that trial is 17 - the number of adjacent pairs of pictures that exist). A Fully Corrected Score for which the normative mean is 50 and the standard deviation (SD) is 10.Higher scores are better cognition. A positive change is improvement in function
Change in Working memory using the List Sorting Test | At baseline, 6 weeks, and 12 weeks
  Working Memory is an ability to store data until the amount stored exceeds one's capacity to hold it. A change will be measured using the List sorting test. This takes 7 minutes. This task requires the participant to recall and sequence different visually and orally presented stimuli. Pictures of different foods and animals are displayed with both an accompanying audio recording and written text that name the item. The participant is asked to say the items back to the examiner in size order from smallest to largest. There are two lists - with unadjusted scores ranging from 0-26. A Fully Corrected Score for which the normative mean is 50 and the standard deviation (SD) is 10.Higher scores are better cognition. A positive change is improvement in function
Change in Processing speed using the Pattern Comparison Test | At baseline, 6 weeks, and 12 weeks
  Processing speed (Pattern Comparison): the amount of data that can be processed within a certain unit of time. It is a measure that reflects mental efficiency. A change will be measured using the Picture Sequence memory test. The test itself takes less than 90 seconds and requires participants to discern whether two side-by-side pictures are the same or not. The test consists of ~130 items or lasts 85 seconds, whichever comes first. Unadjusted scores range from 0-130. A Fully Corrected Score for which the normative mean is 50 and the standard deviation (SD) is 10. Higher Scores are consistent with higher processing speed. Higher scores are better cognition. A positive change is improvement in function
Change in caloric intake | At baseline, 6 weeks, and 12 weeks
  Using the Automated Self-Administered 24-hour Dietary Assessment, we will measure caloric intake per day. Change measured in the difference between calories per day at baseline to follow-up assessment. This is an automated food recall that assess caloric intake. A change in caloric intake will be reported in kcal per day. Reduction in caloric input suggests reduced calorie intake.
Changes in total cholesterol blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in total cholesterol from baseline as milligrams per deciliter (mg/dL). The Mayo Clinic reference range for total cholesterol is less than 200 milligrams per deciliter (mg/dL). Cholesterol is a lipid that is synthesized in most tissues and actively absorbed from the diet. There is a strong association between serum cholesterol concentrations and cardiovascular disease. A reduction will represent an improvement in total cholesterol
Changes in low density lipoprotein blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in low density lipoprotein from baseline as milligrams per deciliter (mg/dL). The Mayo Clinic reference range for low density lipoprotein is less than 100 milligrams per deciliter (mg/dL). Lipoprotein cholesterol measurements are essential in managing risk for atherosclerotic cardiovascular disease (ASCVD). A reduction will represent an improvement in low density lipoprotein cholesterol
Changes in triglycerides blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in triglycerides from baseline as milligrams per deciliter (mg/dL). The Mayo Clinic reference range for triglycerides is less than 150 milligrams per deciliter (mg/dL). Elevated triglycerides are often associated with reduced HDL-C, insulin resistance, hypertension, fatty liver disease, and increased waist circumference. A reduction will represent an improvement in triglycerides
Change in high density lipoprotein blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in high density lipoprotein from baseline as milligrams per deciliter (mg/dL). The Mayo Clinic reference range for high density lipoprotein is greater than or equal to 40 milligrams per deciliter (mg/dL) in males and 50 milligrams per deciliter (mg/dL) for females. Lipoprotein cholesterol measurements are essential in managing risk for atherosclerotic cardiovascular disease (ASCVD). A reduction will represent a worsening in high density lipoprotein cholesterol
Change in C-reactive protein blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in C-reactive protein from baseline as milligrams per liter (mg/L). The Mayo Clinic reference range for C-reactive protein is less than 5 milligrams per liter (mg/L). Measuring changes in the concentration of C-reactive protein (CRP) provides useful diagnostic information about the level of acuity and severity of a disease. It also allows judgments about the disease genesis. A reduction will represent an improvement in c-reactive protein and inflammation
Change in Tumor Necrosis Factor- alpha (TNF-a) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in TNF-a from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for TNF-a is less than 5.6 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders, or may be used for research purposes. A reduction will represent an improvement in tumor necrosis factor alpha and inflammation
Change in Interleukin 1 beta (IL-1-beta) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in IL-1 beta from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for IL-1 beta is less than 6.7 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders, or may be used for research purposes. A reduction will represent an improvement in IL-1 beta and inflammation
Change in Interleukin 6 (IL6) blood levels from baseline | At baseline and 12 weeks
  Measures the change in IL6 from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for IL6 is less than 6.4 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders, or may be used for research purposes. A reduction will represent an improvement in IL-6 and inflammation
Change in stool alpha-diversity levels from baseline | At baseline and 12 weeks
  Change in alpha-diversity from stool collection at baseline. stool 16S Ribosomal ribonucleic acid (rRNA) sequence data processing will yield measures of alpha-diversity and abundances (counts) of distinct taxa (to the genus level). A positive (increase) represents an increase in diversity
Change in serum sample from baseline | At baseline and 12 weeks
  Characterization of response phenotypes to the intervention and the factors associated with inter-individual variability in those responses using bioinformatic identification, and characterization of interactions for future predictive studies. The team will collect a blood sample at baseline (0-weeks) and follow up (12-weeks) to conduct an untargeted metabolomic analysis to demonstrate potential peaks of protein within the blood reported in mg/dL. An untargeted analysis is a process of discovery science where a priori there are no prespecified metabolites but are discovered based on the results of the study.
Change in 30-second sit-to-stand from baseline | At baseline, 6 weeks, and 12 weeks
  The 30-second sit-to-stand test is administered using a folding chair without arms and involves recording the number of stands from a seated position a person can complete in 30 seconds. Change in 30-s sit-to-stand in repetitions over time will be reported from baseline to 12-weeks. An improvement in repetitions will represent an improvement of physical function. Minimal clinically significant change is 2.3 repetitions.
Change in grip strength from baseline | At baseline, 6 weeks, and 12 weeks
  Using a Jamar dynamometer, change in participant's maximal grip strength measurement in kilograms from baseline. Absolute change in grip strength in kilograms over time will be reported from baseline to 12-weeks. An increase in kilograms represented on the device will represent an improvement of physical function. Scale: healthy women aged 70-79 years is 1.13 meters per second (m/s) and for men 1.26 m/s. For women and men aged 80-99 the values are 0.94 meters per second (m/s) and 0.97 meters per second (m/s), respectively.
Change in gait speed from baseline | At baseline, 6 weeks, and 12 weeks
  Gait speed (measured in meters/second or m/s) measures how long it takes a person to travel a given distance. Gait Speed is measured using the time in seconds it takes a participant to complete a 4 meter course while walking at a usual pace. Gait speed is measured as distance (meters) ÷ time (seconds). An absolute change in gait speed will be the difference from follow-up measures and baseline. An improvement in gait speed represents an improvement in physical function. Units are meters/second. Scale: healthy women aged 70-79 years is 1.13 meters per second (m/s) and for men 1.26 m/s. For women and men aged 80-99 the values are 0.94 meters per second (m/s) and 0.97 meters per second (m/s), respectively.
Change in 400-meter walk time from baseline | At baseline, 6 weeks, and 12 weeks
  The 400-meter walk test, measured as time (in seconds) to complete the test. The 400-meter walk will be used to measure cardiorespiratory fitness (CRF) during which individuals will be asked to walk continuously for 400 meters on a flat, indoor surface around cones (separated by at least 20 feet). An absolute change in 400-meter walk time will be the difference from follow-up measures and baseline. An improvement in 400-m walk represents an improvement in aerobic function. Units are meters. A clinically important differences is 34m.
Change in Fat Mass | At baseline and 12 weeks
  An MRI-based measure of body composition consisting of fat mass. This will be measured as volume in mL based on fat mass (adipose) volume of the entire body. A change in Fat Mass over time from baseline to 12-weeks. A reduction in fat mass volume is suggestive of improvements in health related outcomes.
Change in Fractional Percentage of Fat Mass | At baseline and 12 weeks
  An MRI-based measure of body composition. Fat Mass (Fractional Percentage) will be measured as volume in % based on fat mass (adipose) volume of the entire body in relation to the total mass. A change in Fat Mass (fractional percentage) over time from baseline to 12-weeks. A reduction in fat mass percentage is suggestive of improvements in health related outcomes.
Change in Fractional Percentage of Lean Mass | At baseline and 12 weeks
  An MRI-based measure of body composition. Lean Mass (Fractional Percentage) will be measured as volume in % based on lean mass (muscle) volume of the entire body in relation to the total mass. A reduction in lean mass percentage is suggestive of worsening of health related outcomes.
Change in Lean Mass Volume | At baseline and 12 weeks
  An MRI-based measure lean mass (muscle) volume of the entire body. A change in Lean Mass over time from baseline to 12-weeks. A reduction in lean mass volume is suggestive of improvements in health related outcomes.
Change in Fractional Percentage Visceral Mass | At baseline and 12 weeks
  An MRI-based measure of body composition consisting of fat mass. This will be measured as volume in mL based on fat mass (adipose) volume of the entire body. A change in Fat Mass (fractional percentage) over time from baseline to 12-weeks. A reduction in fat mass volume is suggestive of improvements in health related outcomes.
Change in Ultrasound Imaging Intensity | At baseline, 6 weeks, and 12 weeks
  An ultrasound-based measure of body composition. This will be measured as echointensity (no units) based on muscle/fat intensity of the quadricep muscle. A change in echointensity over time from baseline to 12-weeks. A reduction in intensity is suggestive of improvements in health related outcomes.
Change in Pittsburgh Fatigability Scale | At baseline, 6 weeks, and 12 weeks
  The 15-item Pittsburgh Fatigability Scale measures perceived fatigue of sedentary, social, lifestyle and physical activities (light-high intensity, 0-50 scale). Cutoff of ≥15 and ≥13 indicate higher physical and mental fatigue that may lead to reduced performance or restricted activity. Higher scores indicate greater perceived physical or mental fatigability. A reduction in the absolute change in score suggests improvements in fatigue.
Change in Patient reported outcomes measurement information systems (PROMIS) General Health | At baseline, 6 weeks, and 12 weeks
  PROMIS General Health gauges physical, mental, and social aspects of health (5-point scale) to record changes in global health at each time point. A mean standardized score for the population is 50; 10 points indicate one standard deviation. Higher scores indicate better health.
Change in Rates of Physical Activity Type | At baseline, 6 weeks, and 12 weeks
  Physical activity will be assessed using the validated 41-item Community Healthy Activities Model Programs (CHAMPS) questionnaire for older adults. The Community Healthy Activities Model Programs (CHAMPS) assesses usual weekly amounts activity levels and types (activity frequency) and their change. Physical activity is classified as type of activity - low, moderate, vigorous. The change in rates of each type of activity will be presented between baseline and 12-weeks.
Change in Metabolic equivalents | At baseline, 6 weeks, and 12 weeks
  The 41-item Community Healthy Activities Model Programs (CHAMPS) will assess metabolic equivalents per week and their changes; scoring is classified as the number of metabolic equivalents. The change in rates of each type of activity will be presented between baseline and 12-weeks. An increase in metabolic equivalents (METS) suggests improvements in physical function and cardiac function.
Change in Caloric Expenditure with Exercise | At baseline, 6 weeks, and 12 weeks
  The 41-item Community Healthy Activities Model Programs (CHAMPS) will assess weekly caloric expenditure and their changes; scoring is classified as the number of calories expended during exercise. The change in rates of each type of activity will be presented between baseline and 12-weeks. Changes in caloric expenditure of activity (light, moderate, vigorous) will be evaluated. Higher changes in caloric expenditure suggests increased activity.
Change in Social Support for Diet | At baseline, 6 weeks, and 12 weeks
  A validated scale (Sallis et al) that assesses friends/family support for engaging in dietary changes. Higher scores indicate higher social support. Each are scored for family and friends separately (range 0-100).
Change in Social support for exercise | At baseline, 6 weeks, and 12 weeks
  A validated scale (Sallis et al) that assesses friends/family support for engaging in dietary exercises. Higher scores indicate higher social support. Each are scored for family and friends separately (range 0-60).
Compliance Rate of b-hydroxymethylbutyrate | Weekly up to 12 weeks
  Participants will complete a weekly paper or electronic diary to document taking their supplement. Compliance will be calculated as a percent (# of pills taken divided by total # of pills that should have been taken) x 100.
Change in hemoglobin A1C blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in hemoglobin a1c from baseline as a percentage. The Mayo Clinic reference range for hemoglobin a1c is less than 5.7%. The A1C test measures what percentage of hemoglobin proteins in your blood are coated with sugar (glycated). There is a strong association between high hemoglobin a1c blood levels and increased risk of diabetes complications. A reduction will represent an improvement in hemoglobin a1c.
Change in very low density lipoprotein blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in very low density lipoprotein from baseline as milligrams per deciliter (mg/dL). Mayo Clinic states that an elevated VLDL cholesterol level is more than 30 milligrams per deciliter. A reduction will represent an improvement in very low density lipoprotein cholesterol.
Change in interleukin 2 (IL-2) receptor serum levels from baseline | At baseline and 12 weeks
  Measures the absolute change in IL-2 receptor levels from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for IL-2 receptor levels is between 175.3 picograms per milliliter (pg/mL) and 858.2 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders.
Change in interferon gamma serum levels from baseline | At baseline and 12 weeks
  Measures the absolute change in interferon gamma serum from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for interferon gamma serum is less than 8.6 picograms per milliliter (pg/mL).

OTHER OUTCOMES:
Change in interleukin 5 (IL-5) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in interleukin 5 serum from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for interleukin 5 serum is equal to or less than 2.1 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders.
Change in interleukin 13 (IL-13) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in interleukin 13 serum from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for interleukin 13 serum is equal to or less than 2.3 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders.
Change in interleukin 2 (IL-2) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in interleukin 2 serum from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for interleukin 2 serum is equal to or less than 2.1 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders.
Change in blood glucose levels from baseline | At baseline and 12 weeks
  Measures the absolute change in glucose levels from baseline as milligrams per deciliter (mg/dL). The Mayo Clinic reference range for glucose levels is between 80 milligrams per deciliter (mg/dL) and 130 milligrams per deciliter (mg/dL) before meals.
Change in non-high density lipoprotein (non-HDL) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in high density lipoprotein from baseline as milligrams per deciliter (mg/dL). The Mayo Clinic reference range for high density lipoprotein is less than 130 milligrams per deciliter (mg/dL). Lipoprotein cholesterol measurements are essential in managing risk for atherosclerotic cardiovascular disease (ASCVD). An increase will represent a worsening in non-high density lipoprotein cholesterol.
Change in interleukin 12 (IL-12) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in interleukin 12 serum from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for interleukin 12 serum is equal to or less than 1.9 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders.
Change in interleukin 4 (IL-4) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in interleukin 4 serum from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for interleukin 4 serum is equal to or less than 2.2 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders.
Change in interleukin 10 (IL-10) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in interleukin 10 serum from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for interleukin 10 serum is equal to or less than 2.8 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders.
Change in interleukin 8 (IL-8) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in interleukin 8 serum from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for interleukin 8 serum is equal to or less than 3.0 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders.
Change in interleukin 17 (IL-17) blood levels from baseline | At baseline and 12 weeks
  Measures the absolute change in interleukin 17 serum from baseline as picograms per milliliter (pg/mL). The Mayo Clinic reference range for interleukin 17 serum is equal to or less than 1.4 picograms per milliliter (pg/mL). Results are used to understand the pathophysiology of immune, infectious, or inflammatory disorders.

CONTACTS AND LOCATIONS:
Overall Officials: John Batsis, MD, AGSF, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No